CLINICAL TRIAL: NCT03708302
Title: Serratus and Parasternal Infrapectoral Block for Breast Surgery. A Randomized Controlled Double Blinded Study to Measure Impact on Time to Hospital Discharge in an Outpatient Setting.
Brief Title: Serratus and Parasternal Infrapectoral Block for Breast Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112488
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Breast Pain; Post-Op Complication
Keywords: breast surgery; serratus plane block; parasternal infrapectoral block; simple mastectomy; oncoplastic reduction mammoplasty
MeSH Terms: conditions — Mastodynia; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): Ultrasound guided unilateral serratus plane block and unilateral parasternal infrapectoral block with 0.5% ropivacaine.
  Interventions: Procedure: Unilateral serratus plane block; Procedure: Unilateral parasternal infrapectoral block
- Control Group (Sham Comparator): Ultrasound guided unilateral serratus plane block and unilateral parasternal infrapectoral block with 0.9% saline.
  Interventions: Procedure: Unilateral serratus plane block; Procedure: Unilateral parasternal infrapectoral block

INTERVENTIONS:
Procedure: Unilateral serratus plane block — Ultrasound guided unilateral serratus plane block will be performed at the level of 4th rib in anterior axillary line. After skin infiltration with 1% lidocaine, 80mm 22G block needle will be inserted at the caudal aspect of the ultrasound probe and advanced in-plane to target the fascial plane directly below the serratus muscle. Once the tip is verified in the correct position, 20mls of 0.5% ropivacaine will be injected in the plane in 5 mls aliquot after aspiration. Ultrasound guided unilateral parasternal infrapectoral plane block will be performed at the level of 4th rib, lateral to the sternum. After skin infiltration with 1% lidocaine, 80mm 22G block needle will be inserted at the caudal aspect of the ultrasound probe and advanced in-plane to target the fascial plane directly below the pectoralis major muscle. Once the tip is verified in the correct position, 20mls of 0.5% ropivacaine will be injected in the plane slowly in 5 ml aliquots after aspiration.
Procedure: Unilateral parasternal infrapectoral block — Ultrasound guided unilateral serratus plane block will be performed at the level of 4th rib in anterior axillary line. After skin infiltration with 1% lidocaine, 80mm 22G block needle will be inserted at the caudal aspect of the ultrasound probe and advanced in-plane to target the fascial plane directly below the serratus muscle. Once the tip is verified in the correct position, 20 mls of 0.9% saline will be injected in the plane in 5 mls aliquot after aspiration.
  Ultrasound guided unilateral parasternal infrapectoral plane block will be performed at the level of 4th rib, lateral to the sterum. After skin infiltration with 1% lidocaine, 80mm 22G block needle will be inserted at the caudal aspect of the ultrasound probe and advanced in-plane to target the fascial plane directly below the pectoralis major muscle. Once the tip is verified in the correct position, 20 mls of 0.9% saline will be injected in the plane slowly in 5 ml aliquots after aspiration.

SUMMARY:
Effective pain control is important following breast surgery as it improves quality of recovery, decreases the risk of chronic pain development and reduction of overall health care cost. Current strategies of pain management for breast surgery include use of opioid medication or addition of regional anesthesia along with general anesthesia. Serratus block and parasternal infrapectoral blocks are newly developed fascial plane blocks that are technically easy to perform, effective and safe based on our daily clinical practice and published evidence. We are comparing the addition of serratus and parasternal infrapectoral nerve block with general anesthesia to a combination of placebo and general anesthesia for breast reduction surgery. We propose that this would result in an improved efficiency resulting in early hospital discharge and improve quality of patient care, following breast reduction surgery.

DETAILED DESCRIPTION:
Study Introduction:

Severe acute postoperative pain affects nearly 60% of breast surgery patients, potentially triggering adverse physiological and psychological responses, increased chronic pain incidence, and elevated healthcare costs. Effective perioperative pain management reduces chronic pain occurrence, improves recovery quality, and enables early hospital discharge, thus reducing overall healthcare expenses. Various analgesic strategies exist, ranging from regional techniques to opioid-based approaches. Combining multimodal analgesia with regional anesthesia offers superior pain control and enhances recovery quality. The chest wall and breast skin receive innervation from intercostal nerves, with branches providing sensory input to different areas. Understanding this innervation pattern is crucial for optimizing analgesic approaches in breast surgery and ensuring comprehensive pain relief across all affected regions.

Regional analgesic techniques offer several advantages over traditional parenteral opioid therapy, including enhanced pain relief, reduced opioid consumption and related side effects, quicker PACU discharge, and lower chronic pain occurrence. Paravertebral analgesia is particularly effective for breast surgery but presents drawbacks that limit its popularity, such as variable sensory distribution, potential epidural spread, failure rates, and serious risks like total spinal anesthesia or pneumothorax. Interfascial block techniques, aided by ultrasound, have gained traction in regional anesthesia. These techniques involve injecting local anesthetic into neuro-fascial planes adjacent to muscles or between muscle layers, facilitating its distribution to nerves. Interfascial blocks offer advantages like ease of performance, increased safety by avoiding direct nerve targeting, fewer injections, and superficial application, reducing risks associated with deeper nerve blocks. Given these benefits and a thorough understanding of thoracic wall anatomy, several interfascial blocks have been developed as alternatives to paravertebral blocks, aiming for equal efficacy with fewer risks, particularly important in the context of day case breast surgeries.

The serratus block for breast surgery:

The Serratus Plane Block, introduced by Blanco in 2013, involves injecting local anesthetic beneath the serratus anterior muscle to target intercostal nerve branches. However, our recent anatomical study revealed that a single midaxillary line injection inadequately covers the entire breast, prompting additional parasternal injections for comprehensive sensory coverage. Despite this refinement, no randomized controlled trial has yet assessed the efficacy of combined serratus and parasternal infrapectoral blocks in breast surgery analgesia.

Questions and Hypothesis:

1. Primary Question:

   Does the addition of serratus block and parasternal infrapectoral nerve block to patients undergoing breast surgery result in improved perioperative patient care resulting in early hospital discharge (breast reduction mammoplasty and simple mastectomy) compared to patients getting wound infiltration with local anesthetic infiltration by surgeon for analgesia?
2. Secondary Questions:

Does the addition of these blocks to general anesthesia result in other benefits such as:

I. Decreased chronic postoperative pain after 3 months, as assessed at 6 month post-surgery follow-up meeting.

II. less acute post-operative pain. III. less intraoperative opioid consumption. IV. less postoperative opioid consumption. V. less incidence of opioid-related side effects such as nausea, vomitus and pruritus.

VI. greater patient satisfaction with their pain relief improved. VII. greater quality of recovery after anesthesia. VIII. shorter phase I (PACU) and phase II (surgical day care, SDC) recovery times).

Trial Design:

This will be a prospective, double-blinded, randomized and controlled trial conducted at St. Joseph's Hospital, London, Ontario. The study will enroll 133 participants undergoing unilateral simple mastectomy or oncoplastic reduction mammoplasty surgery under general anesthesia. After obtaining written informed consent from eligible patients, study participants will be randomly assigned to one of two groups:

1. Study Group:

   Participants will receive preoperative ultrasound-guided unilateral serratus block with 20 ml of 0.5% ropivacaine on each injection at anterior axillary line at 4th rib and unilateral ultrasound guided parasternal infrapectoral block at the level of 4th with 20ml of 0.5% ropivacaine on each injection, at the surgical site, 15 minutes prior to receiving general anesthesia for the surgery. Patients in the study group will also receive sham injection of saline as infiltration by the surgeon near the conclusion of surgery (40 ml of saline).
2. Control group:

Before general anesthesia, participants will receive a preoperative "placebo injection" of 40 mls of saline instead of ropivacaine for unilateral serratus and parasternal infrapectoral nerve block on the surgical site. Patients will then receive 40 ml of 0.5% ropivacaine as injected by the surgeon as infiltration near the conclusion of surgery.

Patient enrollment and consent:

Patients will be approached for participation in this study when they present for their surgical consultation in the Breast Surgical Clinic or at the surgeon's clinic by the surgical team. They will be provided with information regarding the study (Introduction Letter and Letter of Information and Consent Form) and if they provide consent to be contacted for further information and eligibility assessment. One of study team members will then contact the patient after a week by telephone and review the study with them. They will have all questions addressed by telephone and if they wish to participate, they will bring their consent form with them on the surgery day (to avoid unnecessary visits to hospital during pandemic) and sign consent with a witness prior to any study intervention. They will have a further opportunity to have any questions answered at this time as well and can decline to participate in the study at any time. The signed consent form will be photocopied and they will be provided with a signed copy of their consent form for their records.

Randomization and Blinding:

Patients will be randomized to one of two groups by a computer-generated sequence. Investigators and participants will both be blinded to patient assignment at the time of randomization as well as throughout treatment and assessment. Randomization information will be kept in sealed individual envelopes that are opaque to light and sequentially numbered. Each envelope will only be opened after informed consent is given, and immediately prior to the commencement of the block procedure. The individual who generates the randomization schedule will not have contact with study patients. Patients who are randomized to the control group will receive equivalent volume of normal saline solutions for the bilateral blocks procedure in contrast to the patients in the intervention group who receive four injections of 20mls of 0.5% Ropivaciane for each injection. This is meant to maintain patient and investigator blinding. The anesthetist(s) performing the block will be blinded to the intervention along with the anesthetists performing the general anesthesia and the surgical team. Importantly, the intraoperative and postoperative opioids will be administered by anesthetists and nurses, respectively, who are blinded to group allocation. Furthermore, the research coordinator collecting all outcome data will also be blinded.

Surgical Interventions:

1. Simple Mastectomy:

   Patients undergoing simple mastectomy (removal of breast gland and skin envelope) without immediate reconstruction are typically booked as same day surgeries, meaning they go home after their surgery on the same day. The skin is incised and elevated off the breast gland at the subcutaneous plane, leaving only enough skin for primary wound closure. The breast gland is elevated off the pectoralis fascia which contributes to the majority of postoperative pain. A drain is typically left into the subcutaneous plane and managed by homecare until the drainage is less than 30 cc/24 hour period (most drains are in place for 5-7 days).
2. Oncoplastic reduction mammoplasty:

Oncoplastic breast reduction mammoplasty is another surgical technique meant as a breast conserving alternative to mastectomy in patients with larger, ptotic breasts in whom up to 60% of the breast is affected by disease and needs to be removed. In these procedures, the area of affected breast gland to be removed is excised while sparing the breast skin envelope, and the remaining gland is elevated off the pectoralis fascia and rotated to fill the defect, creating essentially a breast reduction pattern, upon which the breast skin is then redraped, creating a smaller breast without defect.

Preoperative Management:

Standard monitoring (ECG, blood pressure and oxygen saturation monitoring) will be applied, an intravenous access will be established and participants will receive midazolam 1-2 mg IV for anxiolysis as required. They will be positioned supine for the block performance. The skin overlying the chest wall will be disinfected using a chlorhexidine solution and a high-frequency linear ultrasound transducer (6-13 MHz, Sonosite M-Turbo) will be covered with a sterile plastic sheath. The block will be performed under strictly aseptic conditions by a staff regional anesthetist, by two regional anesthesiologists specialized to perform this nerve block.

Intraoperative Management:

All subjects will receive a standardized general anesthesia with a laryngeal mask airway or endotracheal intubation depending on the anesthesiologist looking after the participant for their surgery. They will receive intravenous induction using standard doses of fentanyl 1-2 mcg/kg, propofol 2-4 mg/kg and rocuronium 0.6mg/kg if needed. Anesthesia will be maintained with desflurane/sevoflurane (end-tidal concentration corresponding to 1-1.3 MAC, age-corrected) in a mixture of room air (50%) and oxygen (50%). Positive pressure ventilation will only be initiated when spontaneous ventilation cannot be maintained (e.g. when muscle relaxant is used). Positive pressure support will be titrated to maintain an end-tidal CO2 value of 30-40 mmHg. As per routine practice, fentanyl 1 mcg/kg, morphine 0.05 - 0.1 mg/kg or hydromorphone 0.0075 - 0.015 mg/kg will be administered to treat hemodynamic increases of more than 25% above pre-induction baseline values. As per routine antiemetic prophylaxis, dexamethasone 0.1mg/kg at the beginning of surgery and ondansetron 4 mg IV will be given 30 min before the anticipated end of surgery and dimenhydrinate (gravol) 0.5 mg/kg will only be reserved as a last-line therapy in PACU for otherwise not controllable PONV.

Postoperative pain management:

As per routine practice, morphine 2 mg IV or hydromorphone 0.4 mg IV every 5 min as needed will be administered to all participants with pain on a Numeric Rating Scale (NRS) ≥ 4 or after participant request. As soon as oral intake is started, participants will also have access to oxycodone 5 mg PO when needed. Upon discharge from hospital, participants will receive a prescription for Tylenol #3 (acetaminophen 300 mg/codeine 30 mg per tablet) 1-2 tablets every 4 h as needed or Percocet® (acetaminophen 325 mg/oxycodone HCl 5 mg per tablet) if intolerant to codeine. Participants will be contacted over the phone the following day inquiring about their quality of recovery based on the (QoR-15) questionnaire and will also be asked about their level of pain based on numerical analogue score, total and cumulative oral analgesic consumed since discharge from the hospital, opioid-related side effects, block-related side effects, and satisfaction with postoperative analgesia at postoperative days one.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-80 years
* ASA I to III (American Society of Anesthesiologists Physical Status Classification System)
* Undergoing unilateral oncoplastic breast reduction mammoplasty, simple mastectomy surgery, or lumpectomy at St. Joseph's Hospital.
* Day surgery procedures

Exclusion Criteria:

* Inability to understand or to provide consent
* Inability or unwillingness to comply with required follow-up assessments
* Psychiatric disorder affecting patient assessment
* Contraindication to regional anesthesia, e.g. coagulopathy
* Allergy to local anesthetic
* Chronic pain and/or chronic use of opioids with a daily use of over 30 mg oxycodone or equivalent per day
* Contraindication to a component of multimodal analgesia
* Preexisting neuropathy with motor or sensory deficits in the area of the anterolateral chest wall
* Infection near injection site
* Pregnancy
* BMI>40
* Complication or adverse events unrelated to the study intervention that precludes evaluation of the primary and secondary outcomes.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is based on female patients coming for breast reduction surgery.
Enrollment: 120 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Time to hospital discharge. | 24 hours postoperative period
  Comparing time to hospital discharge; the total time being 'admission to postoperative Care Unit after surgery till discharge home.' this will be measured in minutes

SECONDARY OUTCOMES:
post operative pain score | 48 hours
  Pain score in admission to phase I recovery (PACU), admission to phase II recovery (day surgery unit), and discharge from day surgery unit.
Cumulative Opioid consumption (in Intravenous Morphine equivalent). | 48 hours
  Total opioid consumption at three time points, intraoperative, PACU stage I and PACU stage II
Duration of Hospital stay in minutes. | 24 hours
  Total duration in PACU stage I and in PACU stage II
Opioid-related side effects requiring treatment. | 48 hours
  nausea, vomitus, pruritus and respiratory depression needing medication for treatment or urgent physician assistance.
Presence/absence of block-related side effects. | 48 hours
  bruising, infection, local anesthetic systemic toxicity, persistent numbness of shoulder weakness
Quality of recovery score (QoR) after anesthesia (at discharge and on Post Operative Day 1) | 48 hours
  questionnaire based quality of recovery score

CONTACTS AND LOCATIONS:
Overall Officials: Abhijit Biswas, MD, Principal Investigator — London Health Sciences Center, Western University, London. Ontario. Canada
Locations (1):
- St. Joseph's Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Plan to publish/ share the aggregate summary of the results instead of individual patient data. Individual patients de - identified results could be shared depending on journal requirement at time of publication.

REFERENCES:
- [Background] Fecho K, Miller NR, Merritt SA, Klauber-Demore N, Hultman CS, Blau WS. Acute and persistent postoperative pain after breast surgery. Pain Med. 2009 May-Jun;10(4):708-15. doi: 10.1111/j.1526-4637.2009.00611.x. Epub 2009 Apr 22. PMID 19453965
- [Background] Joshi GP, Ogunnaike BO. Consequences of inadequate postoperative pain relief and chronic persistent postoperative pain. Anesthesiol Clin North Am. 2005 Mar;23(1):21-36. doi: 10.1016/j.atc.2004.11.013. PMID 15763409
- [Background] Sinatra R. Causes and consequences of inadequate management of acute pain. Pain Med. 2010 Dec;11(12):1859-71. doi: 10.1111/j.1526-4637.2010.00983.x. Epub 2010 Oct 28. PMID 21040438
- [Background] Carpenter JS, Andrykowski MA, Sloan P, Cunningham L, Cordova MJ, Studts JL, McGrath PC, Sloan D, Kenady DE. Postmastectomy/postlumpectomy pain in breast cancer survivors. J Clin Epidemiol. 1998 Dec;51(12):1285-92. doi: 10.1016/s0895-4356(98)00121-8. PMID 10086821
- [Background] Tasmuth T, Blomqvist C, Kalso E. Chronic post-treatment symptoms in patients with breast cancer operated in different surgical units. Eur J Surg Oncol. 1999 Feb;25(1):38-43. doi: 10.1053/ejso.1998.0597. PMID 10188853
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Background] Johansen A, Romundstad L, Nielsen CS, Schirmer H, Stubhaug A. Persistent postsurgical pain in a general population: prevalence and predictors in the Tromso study. Pain. 2012 Jul;153(7):1390-1396. doi: 10.1016/j.pain.2012.02.018. Epub 2012 Mar 24. PMID 22445291
- [Background] Jaspars JJ, Posma AN, van Immerseel AA, Gittenberger-de Groot AC. The cutaneous innervation of the female breast and nipple-areola complex: implications for surgery. Br J Plast Surg. 1997 Jun;50(4):249-59. doi: 10.1016/s0007-1226(97)91155-3. PMID 9215081
- [Background] Nasu H, Yamaguchi K, Nimura A, Akita K. An anatomic study of structure and innervation of the serratus anterior muscle. Surg Radiol Anat. 2012 Dec;34(10):921-8. doi: 10.1007/s00276-012-0984-1. Epub 2012 May 26. PMID 22638721
- [Background] Hamada J, Igarashi E, Akita K, Mochizuki T. A cadaveric study of the serratus anterior muscle and the long thoracic nerve. J Shoulder Elbow Surg. 2008 Sep-Oct;17(5):790-4. doi: 10.1016/j.jse.2008.02.009. Epub 2008 Jun 30. PMID 18586531
- [Background] Yeh CC, Yu JC, Wu CT, Ho ST, Chang TM, Wong CS. Thoracic epidural anesthesia for pain relief and postoperation recovery with modified radical mastectomy. World J Surg. 1999 Mar;23(3):256-60; discussion 260-1. doi: 10.1007/pl00013180. PMID 9933696
- [Background] Doss NW, Ipe J, Crimi T, Rajpal S, Cohen S, Fogler RJ, Michael R, Gintautas J. Continuous thoracic epidural anesthesia with 0.2% ropivacaine versus general anesthesia for perioperative management of modified radical mastectomy. Anesth Analg. 2001 Jun;92(6):1552-7. doi: 10.1097/00000539-200106000-00041. PMID 11375845
- [Background] Belzarena SD. Comparative study between thoracic epidural block and general anesthesia for oncologic mastectomy. Rev Bras Anestesiol. 2008 Nov-Dec;58(6):561-8. doi: 10.1590/s0034-70942008000600001. English, Portuguese. PMID 19082403
- [Background] Naja MZ, Ziade MF, Lonnqvist PA. Nerve-stimulator guided paravertebral blockade vs. general anaesthesia for breast surgery: a prospective randomized trial. Eur J Anaesthesiol. 2003 Nov;20(11):897-903. doi: 10.1017/s0265021503001443. PMID 14649342
- [Background] Schnabel A, Reichl SU, Kranke P, Pogatzki-Zahn EM, Zahn PK. Efficacy and safety of paravertebral blocks in breast surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2010 Dec;105(6):842-52. doi: 10.1093/bja/aeq265. Epub 2010 Oct 14. PMID 20947592
- [Background] Tahiri Y, Tran DQ, Bouteaud J, Xu L, Lalonde D, Luc M, Nikolis A. General anaesthesia versus thoracic paravertebral block for breast surgery: a meta-analysis. J Plast Reconstr Aesthet Surg. 2011 Oct;64(10):1261-9. doi: 10.1016/j.bjps.2011.03.025. Epub 2011 Apr 12. PMID 21486711
- [Background] Abdallah FW, Morgan PJ, Cil T, McNaught A, Escallon JM, Semple JL, Wu W, Chan VW. Ultrasound-guided multilevel paravertebral blocks and total intravenous anesthesia improve the quality of recovery after ambulatory breast tumor resection. Anesthesiology. 2014 Mar;120(3):703-13. doi: 10.1097/ALN.0000436117.52143.bc. PMID 24071616
- [Background] Marhofer D, Marhofer P, Kettner SC, Fleischmann E, Prayer D, Schernthaner M, Lackner E, Willschke H, Schwetz P, Zeitlinger M. Magnetic resonance imaging analysis of the spread of local anesthetic solution after ultrasound-guided lateral thoracic paravertebral blockade: a volunteer study. Anesthesiology. 2013 May;118(5):1106-12. doi: 10.1097/ALN.0b013e318289465f. PMID 23442752
- [Background] Naja ZM, El-Rajab M, Al-Tannir MA, Ziade FM, Tayara K, Younes F, Lonnqvist PA. Thoracic paravertebral block: influence of the number of injections. Reg Anesth Pain Med. 2006 May-Jun;31(3):196-201. doi: 10.1016/j.rapm.2005.12.004. PMID 16701182
- [Background] Purcell-Jones G, Pither CE, Justins DM. Paravertebral somatic nerve block: a clinical, radiographic, and computed tomographic study in chronic pain patients. Anesth Analg. 1989 Jan;68(1):32-9. PMID 2910135
- [Background] Lonnqvist PA, MacKenzie J, Soni AK, Conacher ID. Paravertebral blockade. Failure rate and complications. Anaesthesia. 1995 Sep;50(9):813-5. doi: 10.1111/j.1365-2044.1995.tb06148.x. PMID 7573876
- [Background] Naja Z, Lonnqvist PA. Somatic paravertebral nerve blockade. Incidence of failed block and complications. Anaesthesia. 2001 Dec;56(12):1184-8. doi: 10.1046/j.1365-2044.2001.02084-2.x. PMID 11736777
- [Background] Klein SM, Bergh A, Steele SM, Georgiade GS, Greengrass RA. Thoracic paravertebral block for breast surgery. Anesth Analg. 2000 Jun;90(6):1402-5. doi: 10.1097/00000539-200006000-00026. PMID 10825328
- [Background] Terheggen MA, Wille F, Borel Rinkes IH, Ionescu TI, Knape JT. Paravertebral blockade for minor breast surgery. Anesth Analg. 2002 Feb;94(2):355-9, table of contents. doi: 10.1097/00000539-200202000-00023. PMID 11812698
- [Background] Coveney E, Weltz CR, Greengrass R, Iglehart JD, Leight GS, Steele SM, Lyerly HK. Use of paravertebral block anesthesia in the surgical management of breast cancer: experience in 156 cases. Ann Surg. 1998 Apr;227(4):496-501. doi: 10.1097/00000658-199804000-00008. PMID 9563536
- [Background] Piccioni F, Colombo J, Fumagalli L, Lassola S, Previtali P, Ammatuna M, Langer M. Inadvertent high central neuraxial block and possible total spinal anaesthesia occurring after nerve stimulation guided thoracic paravertebral block. Anaesth Intensive Care. 2014 Mar;42(2):270-1. No abstract available. PMID 24580402
- [Background] Abdallah FW, Chan VW, Brull R. Transversus abdominis plane block: a systematic review. Reg Anesth Pain Med. 2012 Mar-Apr;37(2):193-209. doi: 10.1097/AAP.0b013e3182429531. PMID 22286518
- [Background] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Lopez-Matamala B, Fajardo M, Estebanez-Montiel B, Blancas R, Alfaro P, Chana M. A new thoracic interfascial plane block as anesthesia for difficult weaning due to ribcage pain in critically ill patients. Med Intensiva. 2014 Oct;38(7):463-5. doi: 10.1016/j.medin.2013.10.005. Epub 2013 Nov 26. No abstract available. PMID 24289954
- [Background] Kunhabdulla NP, Agarwal A, Gaur A, Gautam SK, Gupta R, Agarwal A. Serratus anterior plane block for multiple rib fractures. Pain Physician. 2014 Jul-Aug;17(4):E553-5. No abstract available. PMID 25054407
- [Result] Biswas A, Luginbuehl I, Szabo E, Caldeira-Kulbakas M, Crawford MW, Everett T. Use of Serratus Plane Block for Repair of Coarctation of Aorta: A Report of 3 Cases. Reg Anesth Pain Med. 2018 Aug;43(6):641-643. doi: 10.1097/AAP.0000000000000801. PMID 29794944
- [Result] Biswas A, Castanov V, Li Z, Perlas A, Kruisselbrink R, Agur A, Chan V. Serratus Plane Block: A Cadaveric Study to Evaluate Optimal Injectate Spread. Reg Anesth Pain Med. 2018 Nov;43(8):854-858. doi: 10.1097/AAP.0000000000000848. PMID 30063656